CLINICAL TRIAL: NCT01553890
Title: Empirical Comparative Study of Variation Blood Level Antibody Vitamin D at SSc Patients Compared Healthy Peoples
Brief Title: Empirical Comparative Study of Variation Blood Level Antibody Vitamin D at Scleroderma (SSc) Patients Compared Healthy Peoples
Acronym: SSc
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: vitamin D and Scleroderma
Record Dates: First submitted 2012-03-05; First posted 2012-03-14 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-01

CONDITIONS: Scleroderma
Keywords: SSc= scleroderma; ICF+ informed consent form; age 18 to 85; healthy
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients diagnosed with scleroderma (Other): patients diagnosed with scleroderma, clinical and lab support
  Interventions: Other: Blood sample
- No disease (Other): Blood sample, venous blood, about 10 ml will be drawn from participants
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — blood sample, venous blood, about 10 ml will be drawn from participants

SUMMARY:
The aim is to find the presence of anti vitamin D antibodies in scleroderma patients and compare with control. A second goal is anti vitamin D levels in serum of scleroderma patients in relation to the clinical manifestations of the disease.

DETAILED DESCRIPTION:
Blood samples from 30 scleroderma patients compared to 30 healthy peoples to reach the target of variation of the blood level vitamin D antibody between this groups

ELIGIBILITY:
Inclusion Criteria:

study group

1. patients with SSc
2. age - 18 years old and older
3. sign ICF control group - healthy people

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-11 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Presence of anti vitamin D antibodies in scleroderma patients compared with control | March 2013 (up to one year)

SECONDARY OUTCOMES:
Anti vitamin D presence and levels in serum in relation to the clinical manifestations of scleroderma | March 2013 (up to one year)